CLINICAL TRIAL: NCT06359730
Title: Incidence, Risk Factors Of Low Anterior Resection Syndrome And Validation Of LARS Score Among Egyptian Patients
Brief Title: Incidence and Risk Factors of Low Anterior Resection Syndrome
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Reham Zakaria Mohamed Ahmed, Principal Investigator, Zagazig University
Other Study IDs: 253/26-March-2024
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer
Keywords: rectal cancer; anterior resection; LARS
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: LARS score questionnaire — LARS score questionnaire is filled by the patient after anterior resection for rectal cancer to study the quality of life

SUMMARY:
Sphincter sparing surgery is oftentimes associated with bowel dysfunction complaints, namely the low anterior resection syndrome (LARS). The LARS questionnaire is widely used to assess this syndrome.

With advances in colorectal surgery, sparing sphincter surgeries are gaining popularity. But symptoms after surgery can affect the quality of life which has psychomotor effects. Low anterior resection syndrome score is a worldwide known questionnaire. Many countries have accredited validation and translation of this questionnaire, but to our knowledge; it is the first time in Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18

  * Diagnosed patients with rectal adenocarcinoma and who received low anterior resection with anastomosis creation or after a minimum 6 months interval after stoma reversal.
  * Tumors of the rectum (2-15 cm) from anal verge

Exclusion Criteria:

* • cognitive dysfunction

  * Having a history of inflammatory bowel disease or any disease with bowel function impairment namely, Crohn's disease, irritable bowel syndrome, ulcerative colitis or others.
  * Age less than 18
  * Metastatic cancer or tumor recurrence
  * Rectal tumors within 2 cm from anal verge( abdominoperineal)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients who had anterior resection surgery for rectal carcinoma
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
age | from 2017 to 2022
  age of the patients in years was recorded from patient records
sex | from 2017 to 2022
  sex of patients was recorded from patient records
medical disease | from 2017 to 2022
  medical disease like diabetes and hypertension was recorded from patient records
site of tumor | from 2017 to 2022
  tumor site was determined in Cm from anal verge by colonoscopy
neoadjuvant therapy | from 2017 to 2022
  history of neoadjuvant therapy before surgery was obtained from patients records
site of anastmosis | from 2017 to 2022
  site of anastmosis after resection was recorded as colo-rectal or colo-anal
type of meso-rectal excision | from 2017 to 2022
  excision of meso-rectum was recorded if it was partial or complete
adjuvant therapy | from 2017 to 2022
  it was recorded from patients records if he\she had chemo- or radiotherapy post-operatively
type of surgery | from 2017 to 2022
  from records; surgery was open or laparoscopic
type of anastmosis | from 2017 to 2022
  type of anastmosis(hand sewen or stappled) obtained from records
LARS score | from 2017 to 2022
  obtained by LARS questionnaire filled by the patient during follow up, it was formed of five questions with different scores on answer choices, interpretaion (0-20) means no LARS, (21- 29) means minor LARS, (30-42) means major LARS

CONTACTS AND LOCATIONS:
Overall Officials: Reham Zakaria, PhD, Principal Investigator — faculty of medicine Zagazig University
Locations (1):
- Zagazig University Hospitals, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD will be shared with other researchers on demand by e- mailing the principle investigator